CLINICAL TRIAL: NCT07369934
Title: Virtual Reality Based Exercise Training Versus Mulligan Mobilization on Shoulder Posture and Function in Subacromial Impingement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohsen Sayed Meselhy, Demonstrator at the Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Virtual reality and Mulligan M
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Subacromial Impingement Syndrome
Keywords: subacromial impingement syndrome; Virtual reality; Mulligan mobilization; shoulder function; shoulder posture
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Active Comparator)
  Interventions: Other: Virtual Reality
- Mulligan mobilization group (Active Comparator)
  Interventions: Other: Mulligan mobilization

INTERVENTIONS:
Other: Virtual Reality — Fully immersive virtual reality mounted headset will be used
  Arms: Virtual reality group
Other: Mulligan mobilization — posterolateral shoulder Mulligan mobilization with movement (MWM) will be used
  Arms: Mulligan mobilization group

SUMMARY:
The study will compare the effect of virtual reality based exercise training versus Mulligan mobilization in addition to exercise therapy added to both groups on shoulder posture and function in subacromial impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be referred from the orthopedic surgeon with a diagnosis of stage II SIS with the following criteria:

  1. Participants ranged in age from 30-50 years old.
  2. Participants are from non-athletes from the general population.
  3. Unilateral shoulder pain that is localized either anteriorly or laterally to the acromion. Pain that occurs or worsens when the affected shoulder is in flexion and/or abduction.
  4. Four of the following should be present in the included patients: Neer impingement test, Hawkins' test, Pain was replicated in the supraspinatus empty-can test, a painful arc of movement from 70° to 120°, and painful greater tuberosity of the humerus.
  5. BMI range 18.5- 29.9 Kg/m².

Exclusion Criteria:

* 1) Patients who, during the previous three months, underwent shoulder physical treatment and/or an acute pain flare.

  2) Patients who have undergone surgeries for tendon repair. 3) Malignancy, epilepsy, pregnant women, and/or systemic conditions like chronic renal or liver failure.

  4) Mini-Mental State Examination test (MMSE) (< 24/30) to exclude cognitive impairment and/or significant vision impairment (if they couldn't read the introduction while wearing the Head Mounted Device (HMD).

  5) Corticosteroid injection during the last three months or used steroids chronically.

  6) Adhesive capsulitis, glenohumeral joint instability, Numbness or tingling of the upper limb, and/or full-thickness tear of the rotator cuff.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during shoulder elevation | pain intensity at the start of session 1 to the end of 1 month of treatment
  It will be measured using the Numerical Pain Rating Scale (NPRS)
Shoulder function | shoulder function at the start of session 1 to the end of 1 month of treatment
  The Shoulder Pain and Disability Index (SPADI) will be used to measure the shoulder function.
Shoulder flexion range of motion | shoulder flexion at the start of session 1 to the end of 1 month of treatment
  The Clinometer Application will be used to measure it.
Shoulder abduction range of motion | shoulder abduction at the start of session 1 to the end of 1 month of treatment
  The Clinometer Application will be used to measure it.
shoulder posture | shoulder posture at the start of session 1 to the end of 1 month of treatment
  Sagittal Shoulder Angle will be used to measure the shoulder posture

SECONDARY OUTCOMES:
Patients' enjoyment | It will be evaluated at the end of the last session (after 1 month)
  A 7-point likert scale will be used to the evaluate the level of the patients' enjoyment at the end of the last session.
patients' adherence to treatment sessions | patients' adherence at the start of session 1 to the end of 1 month of treatment
  patients' numbers of attended sessions will be calculated at the end of 1 month of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy Youssed, Professor Doctor, Study Chair — Cairo University; Afaf M Tahoon, lecturer, Study Director — Cairo University; Mohamed A Kotb, Assistant professor, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steiner, B., Elgert, L., Saalfeld, B., & Wolf, K. H. (2020). Gamification in rehabilitation of patients with musculoskeletal diseases of the shoulder: scoping review. JMIR serious games, 8(3), e19914. https://doi.org/10.2196/19914
- [Background] Smith, J., & Doe, A. (2023). Virtual embodiment for improving range of motion in patients with movement-related shoulder pain: An experimental study. Journal of Rehabilitation Science, 45(2), 123-134.
- [Background] Lin, H. T., Li, Y. I., Hu, W. P., Huang, C. C., & Du, Y. C. (2019). A scoping review of the efficacy of virtual reality and exergaming on patients of musculoskeletal system disorder. Journal of clinical medicine, 8(6), 791. https://doi.org/10.3390/jcm8060791
- [Background] Hoyek, N., Di Rienzo, F., Collet, C., Hoyek, F., & Guillot, A. (2014). The therapeutic role of motor imagery on the functional rehabilitation of a stage II shoulder impingement syndrome. Disability and rehabilitation, 36(13), 1113-1119.
- [Background] Consigliere, P., Haddo, O., Levy, O., & Sforza, G. (2018). Subacromial impingement syndrome: management challenges. Orthopedic research and reviews, 83-91. https://doi.org/10.2147/ORR.S157864
- [Background] Coja, D. M., Onu, I., Onu, A., Iordan, D. A., Gheorghiu, G., Ene-Voiculescu, V., & Talaghir, L. G. (2024). The Use of Virtual Reality-Assisted Therapy to Improve Shoulder function in Subacromial Impingement Syndrome: a Randomised Controlled Trial. BRAIN. Broad Research in Artificial Intelligence and Neuroscience, 15(4), 11-26. http://dx.doi.org/10.70594/brain/15.4/2
- [Background] Chaplin, E., Karatzios, C., & Benaim, C. (2023, December). Clinical applications of virtual reality in musculoskeletal rehabilitation: A scoping review. In Healthcare (Vol. 11, No. 24, p. 3178). MDPI. https://doi.org/10.3390/healthcare11243178
- [Background] Álvarez de la Campa Crespo, M., Donegan, T., Amestoy-Alonso, B., Just, A., Combalía, A., & Sanchez-Vives, M. V. (2023). Virtual embodiment for improving range of motion in patients with movement-related shoulder pain: An experimental study. Journal of Orthopaedic Surgery and Research, 18(1), 729. https://doi.org/10.1186/s13018-023-04158-w
- [Result] Özlü, A., Üstündağ, S., Bulut Özkaya, D., & Menekşeoğlu, A. K. (2024). Effect of exergame on pain, function, and quality of life in shoulder impingement syndrome: a prospective randomized controlled study. Games for Health Journal, 13(2), 109-119. https://doi.org/10.1089/g4h.2023.0108
- [Result] Gumaa, M., & Rehan Youssef, A. (2019). Is virtual reality effective in orthopedic rehabilitation? A systematic review and meta-analysis. Physical therapy, 99(10), 1304-1325. https://doi.org/10.1093/ptj/pzz093
- [Result] Dias, D., Neto, M. G., Sales, S. D. S. R., Cavalcante, B. D. S., Torrierri Jr, P., Roever, L., & Araujo, R. P. C. D. (2023). Effect of mobilization with Movement on Pain, disability, and Range of Motion in patients with Shoulder Pain and Movement Impairment: a systematic review and Meta-analysis. Journal of Clinical Medicine, 12(23), 7416. https://doi.org/10.3390/jcm12237416
- [Result] Delgado-Gil, J. A., Prado-Robles, E., Rodrigues-de-Souza, D. P., Cleland, J. A., Fernández-de-las-Peñas, C., & Alburquerque-Sendín, F. (2015). Effects of mobilization with movement on pain and range of motion in patients with unilateral shoulder impingement syndrome: a randomized controlled trial. Journal of manipulative and physiological therapeutics, 38(4), 245-252. https://doi.org/10.1016/j.jmpt.2014.12.008